CLINICAL TRIAL: NCT02147808
Title: A Phase 1, Open-Label, Single-Center, 2-Period, Single-Sequence Drug-Drug Interaction Study to Evaluate the Effects of Multiple-Dose Telotristat Etiprate on the Pharmacokinetics of Single-Dose Midazolam, a Sensitive P450-3A4 Substrate, in Healthy Male and Female Subjects
Brief Title: A Open-Label Drug-Drug Interaction Study of Telotristat Etiprate and Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LX1606.1-108-NRM; LX1606.108 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2014-05-19; First posted 2014-05-28 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Drug Interactions
MeSH Terms: interventions — telotristat; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All subjects will receive a single oral midazolam dose on Day 1 while fasting. Days 2 to 4 will be Washout days. On Day 5, subjects will begin a 5-day regimen of telotristat etiprate. On Day 9, subjects will receive a morning dose of telotristat etiprate with a single dose of midazolam while fasting.
  Interventions: Drug: Telotristat etiprate; Drug: Midazolam

INTERVENTIONS:
Drug: Telotristat etiprate — All subjects will receive two 250 mg telotristat etiprate tablets three times daily.
Drug: Midazolam — All subjects will receive 3 mg (1.5 mL oral syrup [2mg/mL]).

SUMMARY:
This study is designed to evaluate the effects of telotristat ethyl on the pharmacokinetics of midazolam in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females ≥18 to ≤55 years of age at Screening.
* Body mass index ≥18.0 to ≤2.0 kg/m^2
* Acceptable vital signs at Screening: Systolic blood pressure = 90-140 mm Hg, Diastolic blood pressure = 50-90 mm Hg, Heart rate = 40-100 beats per minute
* Willingness to adhere to the restrictions outlines in the protocol
* Able to comprehend and sign the informed consent form.

Exclusion Criteria:

* Presence of any clinically significant physical, laboratory, or ECG finding that may interfere with the study in the opinion of the Investigator
* Use of any medications, herbal tea, energy drink, herbal products, or supplements
* Receipt of any investigational agent or study drug within 30 days or 5 half-lives of study start
* Receipt of any protein- or antibody-based therapeutic agent within 3 months of study start
* Prior exposure to telotristat etiprate
* Use of tobacco, smoking cessation products, or nicotine products within 3 months of study start
* History of major surgery within 6 months of study start
* History of acute narrow angle glaucoma
* History of renal disease, or significantly abnormal glomerular filtration rate (<90 mL/min as calculated using the Cockcroft-Gault equation) at Screening
* History of hepatic disease, or significantly abnormal liver function tests
* History of any clinically significant psychiatric, renal, hepatic, pancreatic, cardiovascular, neurological, endocrinologic, hematological, or GI abnormality
* History of any active infection within 14 days prior to first dosing
* History of alcohol or substance abuse within 2 years prior to Screening
* Positive hepatitis panel (including hepatitis B surface antigen and hepatitis C virus antibody) or positive human immunodeficiency virus antibody screens
* Concurrent conditions that could interfere with safety and/or tolerability measurements
* Donation or loss of >500 mL of blood or blood product within 3 months
* Women who are breastfeeding or are planning to become pregnant during the study
* Positive serum pregnancy test (females only)
* Positive urine screen for selected drugs of abuse and cotinine
* Consumption of alcohol within 48 hours prior to study start
* Consumption of caffeine- and/or xanthine-containing products
* Consumption of grapefruit, Seville oranges, and grapefruit- or Seville orange-containing products within 72 hours prior to study start
* Unable or unwilling to communicate or cooperate with the Investigator for any reason
* Use of any drugs or substances that are known to be substrates, inducers, or inhibitors of CYP3A4 within 30 days prior to the first dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Midazolam plasma concentration in combination with steady state telotristat etiprate | Day 9

SECONDARY OUTCOMES:
Number of treatment emergent adverse events | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Madison, Wisconsin, United States